CLINICAL TRIAL: NCT02413190
Title: Bone Health in Facioscapulohumeral Muscular Dystrophy: A Cross-sectional Study
Brief Title: Bone Health in Facioscapulohumeral Muscular Dystrophy
Acronym: FSHD
Status: Completed | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Concord Hospital (Other); FSHD Global Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00031738
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-02

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a cross-sectional single visit study to determine bone health in individuals with FSHD.

DETAILED DESCRIPTION:
Bone health will be assessed using 1) a DEXA scan to measure bone mineral density and lean body mass, and 2) blood tests of biomarkers of bone resorption and formation. These procedures will be correlated to measures of muscle strength testing and timed function tests to determine fracture risk in FSHD individuals considering age, gender, muscle strength and FSHD allele size.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of FSHD including chromosome 4 deletion and haplotype
* Age > 18 years
* Ability to provide written informed consent for participation in the study
* Ability to participate in the DEXA scan

Exclusion Criteria:

* Unwillingness or inability to comply with the requirements of this protocol (in the opinion of the PI) including, but not limited to, the presence of any condition (physical, mental or social) that precludes the participant from comfortably and safely obtaining a DEXA scan, phlebotomy, or neurological examination

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of individuals with Facioscapulohumeral Muscular Dystrophy.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Kennedy Krieger Institute, Johns Hopkins School of Medicine, Baltimore, Maryland, United States
- Concord Hospital Neurology Department, Hospital Road, Concord NSW 2139, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FSHD: 94 subjects
Period: Overall Study
Arm/Group | FSHD
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- FSHD: 94 subjects with genetically confirmed FSHD1
Arm/Group | FSHD
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (51.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 88
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48
  Australia | 46

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density in FSHD
Description: To determine if bone mineral density is reduced in individuals with FSHD compared to normative data of individuals of the same age and gender without FSHD.The Bone Mineral Density Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population
Time Frame: Single visit
Population: Z score: Higher numbers represent higher bone mineral density.
Measure: Mean (Full Range); unit: z-score
Arm/Group | FSHD
Number analyzed (Participants) | 94
z-score | -0.4 [-4.0 to 3.0]

ADVERSE EVENTS:
Groups:
- FSHD: All subjects with a confirmed FSHD allele
Arm/Group | FSHD
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No